CLINICAL TRIAL: NCT04081636
Title: Prospective, Randomized Study Comparing Transperineal and Transrectal Prostate Biopsy Efficacy and Complications (ProBE-PC Trial)
Brief Title: Prostate Biopsy, Transrectal vs. Transperineal: Efficacy and Complications
Acronym: ProBE-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Badar M. Mian, Professor of Surgery, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 5479
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; PSA; Infection
Keywords: Prostate biopsy; PSA; infection; bleeding
MeSH Terms: conditions — Prostatic Neoplasms; Infections; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to either trans-rectal needle biopsy (TR-Bx) or Trans-perineal biopsy (TP-Bx) of the prostate.
  Both arms, either with or without MRI guided biopsy
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Systematic Transrectal biopsy (TR-Bx) (Active Comparator): Ultrasound guided; needle inserted through the rectum to reach the prostate
  Interventions: Procedure: Systematic Transrectal biopsy (TR-Bx)
- Targeted Transrectal biopsy (TR-Bx) (Active Comparator): MRI-guided; needle inserted through the rectum to reach the prostate
  Interventions: Procedure: Targeted Transrectal biopsy (TR-Bx)
- Systematic Transperineal biopsy (TP-Bx) (Experimental): Ultrasound guided; needle inserted directly through the skin to reach the prostate
  Interventions: Procedure: Systematic Transperineal biopsy (TP-Bx)
- Targeted Transperineal biopsy (TP-Bx) (Experimental): MRI-guided; needle inserted directly through the skin to reach the prostate
  Interventions: Procedure: Targeted Transperineal biopsy (TP-Bx)

INTERVENTIONS:
Procedure: Systematic Transrectal biopsy (TR-Bx) — Through the rectum
  Other Names: ultrasound guided
  Arms: Systematic Transrectal biopsy (TR-Bx)
Procedure: Targeted Transrectal biopsy (TR-Bx) — Through the rectum
  Other Names: MRI guided
  Arms: Targeted Transrectal biopsy (TR-Bx)
Procedure: Systematic Transperineal biopsy (TP-Bx) — Through the perineal skin
  Other Names: ultrasound guided
  Arms: Systematic Transperineal biopsy (TP-Bx)
Procedure: Targeted Transperineal biopsy (TP-Bx) — Through the perineal skin
  Other Names: MRI guided
  Arms: Targeted Transperineal biopsy (TP-Bx)

SUMMARY:
This study evaluates the difference between 2 prostate biopsy methods, transrectal (through the rectal wall) and transperineal (through the skin) needle biopsy.

Men who are in need of prostate biopsy due to clinical suspicions of prostate cancer will be randomly assigned (1:1) to either transrectal or transperineal approach.

This research study will scientifically determine if one biopsy method is better than the other in reducing complications and improving cancer detection.

DETAILED DESCRIPTION:
There are two ways to take biopsy (tissue) samples from the prostate. The more commonly used method is trans-rectal needle biopsy of the prostate (TR-Bx) with a needle inserted through a probe in the rectum to reach the prostate.

TR-Bx is usually performed in the office, using local anesthesia, and often using a targeted biopsy approach using MRI/ultrasound fusion technique.

Trans-perineal biopsy (TP-Bx) with a needle inserted directly through the skin to reach the prostate.

Typically, TP-BX is performed in the outpatient surgical setting due significant pain associated with the procedure, requiring the use anesthesia and/or sedation.

TP-Bx. procedure is very uncommon in the USA and is often performed using ultrasound alone (less accurate), without the benefit of MRI guided targeted biopsy.

Now, with the availability of new devices, we are able to perform both TR-Bx and TP-Bx using MRI/ultrasound fusion guided targeted approach, in the office setting, using local anesthesia alone.

With the TR-Bx, there has been increasing risk of infection related complications, sepsis and hospital admissions.

The newer approach of biopsy TP-Bx may cause fewer infections and may have a higher accuracy of finding cancer.

Using validated questionnaires such as IIEF-6, IPSS and TRUS-BxQ, this randomized study of TR-BX and TP-Bx will address these questions:

* Differences in the risk of infectious complications
* Differences in the overall cancer detection rate and the high-grade cancer detection rate
* Differences in the hemorrhagic and urinary side effects
* Tolerability of both techniques with local anesthesia alone
* Difference in the results of of MRI/US fusion targeted biopsy
* Differences in the cost of the procedures

ELIGIBILITY:
Inclusion Criteria:

* All patients who are scheduled to undergo prostate biopsy for suspected prostate cancer as part of their regular medical care
* Either with or without an MRI

Exclusion Criteria:

* Patients with no access to rectum (due to previous rectal surgery)
* Any abnormalities of the perineal skin (e.g. infection)
* Patients whose procedure requires sedation or general anesthesia

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of infectious complications | 30 days
  Whether or not patient had an infection after the biopsy
Clinically significant cancer detection rate | 14 days
  The rate of grade group 2 prostate cancer detected in each study arm

SECONDARY OUTCOMES:
Rate of Bleeding complications | 30 days
  The type of bleeding and its severity (blood in urine or stool)
Tolerability under local anesthesia | 30 days
  Pain scores; Need for additional analgesia
Patient reported urinary function measures using IPSS questionaire | 30 days
  International Prostate Symptoms Score (IPSS) to measure urinary function
Cost of the procedures | 30 days
  Differences in the actual cost of the procedures (including supplies, time)
Patient reported sexual function measures using IIEF questionaire | 30 days
  International Index of Erectile Function (IIEF) to measure sexual dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Badar M Mian, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical College, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi YH, Kang MY, Sung HH, Jeon HG, Chang Jeong B, Seo SI, Jeon SS, Kim CK, Park BK, Lee HM. Comparison of Cancer Detection Rates Between TRUS-Guided Biopsy and MRI-Targeted Biopsy According to PSA Level in Biopsy-Naive Patients: A Propensity Score Matching Analysis. Clin Genitourin Cancer. 2019 Feb;17(1):e19-e25. doi: 10.1016/j.clgc.2018.09.007. Epub 2018 Sep 13. PMID 30415878
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Moldovan PC, Van den Broeck T, Sylvester R, Marconi L, Bellmunt J, van den Bergh RCN, Bolla M, Briers E, Cumberbatch MG, Fossati N, Gross T, Henry AM, Joniau S, van der Kwast TH, Matveev VB, van der Poel HG, De Santis M, Schoots IG, Wiegel T, Yuan CY, Cornford P, Mottet N, Lam TB, Rouviere O. What Is the Negative Predictive Value of Multiparametric Magnetic Resonance Imaging in Excluding Prostate Cancer at Biopsy? A Systematic Review and Meta-analysis from the European Association of Urology Prostate Cancer Guidelines Panel. Eur Urol. 2017 Aug;72(2):250-266. doi: 10.1016/j.eururo.2017.02.026. Epub 2017 Mar 21. PMID 28336078
- [Background] Wu YP, Li XD, Ke ZB, Chen SH, Chen PZ, Wei Y, Huang JB, Sun XL, Xue XY, Zheng QS, Xu N. Risk factors for infectious complications following transrectal ultrasound-guided prostate biopsy. Infect Drug Resist. 2018 Sep 17;11:1491-1497. doi: 10.2147/IDR.S171162. eCollection 2018. PMID 30271182
- [Background] Borghesi M, Ahmed H, Nam R, Schaeffer E, Schiavina R, Taneja S, Weidner W, Loeb S. Complications After Systematic, Random, and Image-guided Prostate Biopsy. Eur Urol. 2017 Mar;71(3):353-365. doi: 10.1016/j.eururo.2016.08.004. Epub 2016 Aug 17. PMID 27543165
- [Background] Liss MA, Ehdaie B, Loeb S, Meng MV, Raman JD, Spears V, Stroup SP. An Update of the American Urological Association White Paper on the Prevention and Treatment of the More Common Complications Related to Prostate Biopsy. J Urol. 2017 Aug;198(2):329-334. doi: 10.1016/j.juro.2017.01.103. Epub 2017 Mar 29. PMID 28363690
- [Background] Saade EA, Suwantarat N, Zabarsky TF, Wilson B, Donskey CJ. Fluoroquinolone-Resistant Escherichia coli Infections After Transrectal Biopsy of the Prostate in the Veterans Affairs Healthcare System. Pathog Immun. 2016;1(2):243-257. doi: 10.20411/pai.v1i2.123. PMID 27774521
- [Background] Xiang J, Yan H, Li J, Wang X, Chen H, Zheng X. Transperineal versus transrectal prostate biopsy in the diagnosis of prostate cancer: a systematic review and meta-analysis. World J Surg Oncol. 2019 Feb 13;17(1):31. doi: 10.1186/s12957-019-1573-0. PMID 30760274
- [Background] Skouteris VM, Crawford ED, Mouraviev V, Arangua P, Metsinis MP, Skouteris M, Zacharopoulos G, Stone NN. Transrectal Ultrasound-guided Versus Transperineal Mapping Prostate Biopsy: Complication Comparison. Rev Urol. 2018;20(1):19-25. doi: 10.3909/riu0785. PMID 29942197
- [Background] Roberts MJ, Bennett HY, Harris PN, Holmes M, Grummet J, Naber K, Wagenlehner FME. Prostate Biopsy-related Infection: A Systematic Review of Risk Factors, Prevention Strategies, and Management Approaches. Urology. 2017 Jun;104:11-21. doi: 10.1016/j.urology.2016.12.011. Epub 2016 Dec 19. PMID 28007492
- [Background] Altok M, Kim B, Patel BB, Shih YT, Ward JF, McRae SE, Chapin BF, Pisters LL, Pettaway CA, Kim J, Demirel HC, Davis JW. Cost and efficacy comparison of five prostate biopsy modalities: a platform for integrating cost into novel-platform comparative research. Prostate Cancer Prostatic Dis. 2018 Nov;21(4):524-532. doi: 10.1038/s41391-018-0056-7. Epub 2018 Jul 9. PMID 29988098
- [Background] Stefanova V, Buckley R, Flax S, Spevack L, Hajek D, Tunis A, Lai E, Loblaw A; Collaborators. Transperineal Prostate Biopsies Using Local Anesthesia: Experience with 1,287 Patients. Prostate Cancer Detection Rate, Complications and Patient Tolerability. J Urol. 2019 Jun;201(6):1121-1126. doi: 10.1097/JU.0000000000000156. PMID 30835607
- [Background] Meyer AR, Joice GA, Schwen ZR, Partin AW, Allaf ME, Gorin MA. Initial Experience Performing In-office Ultrasound-guided Transperineal Prostate Biopsy Under Local Anesthesia Using the PrecisionPoint Transperineal Access System. Urology. 2018 May;115:8-13. doi: 10.1016/j.urology.2018.01.021. Epub 2018 Feb 1. PMID 29409845
- [Derived] Mian BM, Feustel PJ, Aziz A, Kaufman RP Jr, Bernstein A, Fisher HAG. Clinically Significant Prostate Cancer Detection Following Transrectal and Transperineal Biopsy: Results of the Prostate Biopsy Efficacy and Complications Randomized Clinical Trial. J Urol. 2024 Jul;212(1):21-31. doi: 10.1097/JU.0000000000003979. Epub 2024 May 3. PMID 38700844